CLINICAL TRIAL: NCT02333084
Title: The Influence Of a Natural Anti-Inflammatory Product On Levels Of Inflammatory Markers In Cases With Osteoarthritis Of Knee
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Physician Recommended Nutriceuticals (Industry)
Collaborators: Rothman Institute Orthopedics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRN 20141
Record Dates: First submitted 2014-10-06; First posted 2015-01-07 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Joint Health Product (Experimental): natural dietary supplement
  Interventions: Dietary Supplement: PRN Joint Health Formula
- Placebo (Placebo Comparator): vegetable oil placebo
  Interventions: Dietary Supplement: placebo
- Combination with Omega-3 (Active Comparator): combination with omega-3 fish oil
  Interventions: Dietary Supplement: PRN Flex Omega Benefits® combination

INTERVENTIONS:
Dietary Supplement: PRN Joint Health Formula
  Arms: Joint Health Product
Dietary Supplement: placebo
  Arms: Placebo
Dietary Supplement: PRN Flex Omega Benefits® combination
  Arms: Combination with Omega-3

SUMMARY:
This is a randomized, placebo controlled study. The first subject is expected to be enrolled in July 2014, and the last subject is expected to complete the study by July 2015. Each subject will be provided with the PRN Joint Comfort Formula, placebo or PRN Flex Omega Benefits® combination depending on randomization (1:1:1 at each site) during the course of the study. Instructions and frequency of use will be determined by the labelling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 90 at the time of informed consent.
* Subjects with symptomatic moderate arthritis of the knee defined as per
* Kellgren-Lawrence grade II or III (Appendix B). Subjects with bilateral arthritis of the knee will also be recruited, but only one knee will be enrolled into the study.
* Ability to walk 50 feet unassisted.
* Lequesne's Functional Index score greater than 7 points

Exclusion Criteria:

* Subjects with systemic inflammatory conditions such as inflammatory bowel disease, psoriasis, eczema, and others
* Subjects with seropositive or sero-negative inflammatory arthritis of the knee such as rheumatoid arthritis or ankylosing spondylitis.
* Subjects taking hormone replacement therapy
* Intra-articular corticosteroid injections 3 weeks prior to enrollment.
* Hypersensitivity to fish oil.
* Hypersensitivity to non-steroidal anti-inflammatory drugs, abnormal liver of kidney function tests, history of peptic ulceration and upper gastrointestinal hemorrhage, congestive heart failure, Hypertension (BP>140/90), cancer and hyperkalemia.
* Major abnormal findings on complete blood count, history of coagulopathies, hematological or neurological disorders.
* High alcohol intake (>2 standard drinks per day). Pregnant, breastfeeding or planning to become pregnant during the study
* Subjects awaiting surgery on the affected knee within three months.
* Consumption of any other vitamins/supplements will be allowed, provided the dose is not increased, and same brand is continued with. Also, the regimen should not contain the same active compounds tested in the PRN Joint health formula product.
* Vitamins/supplements cannot be introduced during a subject's participation in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Human Inflammation Multi analyte profile (MAP) v1.0 in Synovial fluid and blood | 12 weeks
  46 different markers of inaflammation will be studies

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 weeks
Pain scores on Visual analog scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Javad Parvizi, MD, Principal Investigator — Rothman Institute
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States